CLINICAL TRIAL: NCT05677763
Title: A Randomised, Placebo-Controlled, 3-Arm, Double-Blind, Multicentre, Phase 4 Study to Assess the Efficacy of OM-85 (Broncho-Vaxom) Short- and Long-Term Treatment vs. Placebo in the Prevention of Respiratory Tract Infections in Children Aged Between 6 Months and 5 Years With Wheezing Lower Respiratory Illness
Brief Title: OM-85 in Paediatric Recurrent Respiratory Tract Infections With Wheezing Lower Respiratory Illness
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: OM Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BV-2020/08; 2024-511581-37-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-14; First posted 2023-01-10 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Tract Infections; Wheezing Lower Respiratory Illness
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BV-12 (Experimental): Subjects will receive OM-85 treatment for 12 consecutive months. (10 days per month)
  Interventions: Drug: OM-85
- BV-3 (Experimental): Subjects will receive OM-85 treatment for 3 consecutive months, followed by matching placebo for 9 consecutive months. (10 days per month)
  Interventions: Drug: OM-85
- Placebo (Placebo Comparator): Subjects will receive matching placebo for 12 consecutive months. (10 days per month)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OM-85 — Subjects will be administered OM-85 3.5 mg capsules by mouth once daily. (10 days per month)
  Arms: BV-12; BV-3
Drug: Placebo — Subjects will be administered Placebo once daily. (10 days per month)
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of OM-85 compared to placebo in reducing the number of respiratory tract infections (RTIs) in children aged between 6 months and 5 years.

DETAILED DESCRIPTION:
This is a Phase 4, randomised, double-blind, placebo-controlled study to assess the efficacy and safety of short- and long-term treatment with OM-85.

The study will consist of screening (up to 20 days before randomisation), Treatment period of 12 months, and an Observational period of 6 months.

The subjects will be randomised in a ratio of 1:1:1 ratio to receive either OM-85 for 12 consecutive months (BV-12 arm), or OM-85 for 3 consecutive months followed by matching placebo for 9 consecutive months (BV-3 arm), or placebo for 12 consecutive months (Placebo arm).

The expected duration of subject participation is 18 months (+20 days).

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender aged between 6 months and 5 years, at Baseline/Randomisation (Visit 2) inclusive.
* For children ≥1 year of age, ≥4 RTIs (as reported by parents or LAR of subject), including ≥2 episodes of wLRIs (including ≥1 triggering hospitalisation or medical visit) within 12 months prior to enrolment.

OR

* For children <1 year of age, ≥2 RTIs (as reported by parents or LAR of subject), including ≥1 episode of wLRIs (including ≥1 triggering hospitalisation or medical visit) within 6 months prior to enrolment.
* Parents or LAR of subject have provided the appropriate written informed consent. Written informed consent must be provided before any study-specific procedures are performed including screening procedures.

Exclusion Criteria:

* Anatomic alterations of the respiratory tract.
* Other chronic respiratory diseases (e.g., tuberculosis, cystic fibrosis).
* Any autoimmune disease.
* HIV infection or any type of congenital or iatrogenic immune deficiency (including IgA deficiency).
* Known severe congenital heart disease.
* Haematologic diseases.
* Liver or kidney failure.
* New-borns before 34 weeks of gestational age.
* Malnutrition as per World Health Organization (WHO) definition.
* Any known neoplasia or malignancy.
* Treatment with the following medications:

  1. Injection or oral administration of steroids within 4 weeks prior to study enrolment.
  2. Previous and/or concomitant immunosuppressants, immunostimulants, or gamma globulins within 6 months prior to study enrolment.
* Previous use within last 6 months of enrolment or ongoing use of bacterial lysates.
* Any major surgery within the last 3 months prior to study enrolment.
* Known allergy or previous intolerance to investigational medicinal products (IMP).
* Any other clinical conditions, that in the opinion of the Investigator, would not allow safe completion of the clinical study.
* Other household members have previously been randomised in this clinical study.
* Subjects' families expected to relocate out of study area within 24 months of the initiation of the study.
* Currently enrolled in or has completed any other investigational device or drug study or receiving other investigational agent(s) within <30 days prior to screening.
* Parents or legally acceptable representative (LAR) who do not have access to internet connection.
* Wheezing documented to be caused by gastroesophageal reflux.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 525 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Rate of respiratory tract infections (RTIs) | 12 Months
  The number of RTIs experienced by a subject during the Treatment period will be assessed.

SECONDARY OUTCOMES:
Rate of wheezing lower respiratory infections (wLRIs) experienced by a subject | 12 Months
  The number of wLRIs experienced by a subject during the Treatment period will be assessed. This is the key secondary endpoint
Rate of wLRIs | 18 Months
  The number of wLRIs experienced by a subject during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Rate of respiratory tract infections (RTIs) | 18 Months
  The number of RTIs experienced by a subject during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Proportion of subjects with recurrent RTIs | 12 Months
  The proportion of subjects experiencing ≥3 RTIs during the first 6 months of treatment, and the number of subjects experiencing ≥4 RTIs during the full 12-month Treatment period will be assessed.
Proportion of subjects with wLRIs | 18 Months
  The proportion of subjects with wLRIs during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Rate of severe wheezing lower respiratory illness (SwLRIs) | 18 Months
  The number of SwLRIs experienced by a subject during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Proportion of subjects with SwLRIs | 18 Months
  The proportion of subjects with SwLRIs during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Time to first, second and third RTI and wLRI | 18 Months
  Time to first, second and third RTI and wLRI will be assessed.
Mean duration in days per RTI | 18 Months
  Mean duration in days per RTI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Mean duration in days per wLRI | 18 Months
  Mean duration in days per wLRI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Number of outpatient medical visits | 18 Months
  Number of outpatient medical visits (hospitalisations, visits to emergency rooms, or to a physician/health care provider) due to an RTI and/or a wLRI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Number of absent days from day-care | 18 Months
  Number of absent days from day-care due to an RTI and/or a wLRI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Number of antibiotic treatments for a respiratory event | 18 Months
  Number of antibiotic treatments for a respiratory event during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Duration of antibiotic treatments for a respiratory event | 18 Months
  Duration of antibiotic treatments for a respiratory event during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Number of systemic corticosteroids, inhaled corticosteroids (ICS) and β2-agonist treatments for a wLRI | 18 Months
  Number of systemic corticosteroids, ICS and β2-agonist treatments for a wLRI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Duration of systemic corticosteroids, ICS and β2-agonist treatments for a wLRI | 18 Months
  Duration of systemic corticosteroids, ICS and β2-agonist treatments for a wLRI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Symptom duration as per the adapted Wisconsin Upper Respiratory Symptom Survey for Kids (WURSS-K) questionnaire | 18 Months
  Symptom duration during the Treatment period, during the Observational period, and during the whole study period will be assessed using WURSS-K questionnaire. Adapted WURSS-K is a valid and reliable illness-specific quality of life instrument that evaluates the impacts of RTIs on children.
Symptom types as per the adapted WURSS-K questionnaire | 18 Months
  Symptom types during the Treatment period, during the Observational period, and during the whole study period will be assessed using WURSS-K questionnaire. Adapted WURSS is a valid and reliable illness-specific quality of life instrument that evaluates the impacts of RTIs on children.
Symptom severity as per the adapted WURSS-K questionnaire | 18 Months
  Symptom severity during the Treatment period, during the Observational period, and during the whole study period will be assessed using WURSS-K questionnaire. Adapted WURSS is a valid and reliable illness-specific quality of life instrument that evaluates the impacts of RTIs on children.
Proportion of subjects who have not used antibiotics as rescue medication for RTI | 18 Months
  The proportion of subjects who have not used antibiotics as rescue medication for RTI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Proportion of subjects who have not been hospitalised for an RTI | 18 Months
  The proportion of subjects who have not been hospitalised for an RTI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Proportion of subjects who have not been administered a systemic corticosteroid for wLRI | 18 Months
  The proportion of subjects who have not been administered a systemic corticosteroid for wLRI during the Treatment period, during the Observational period, and during the whole study period will be assessed.
Proportion of subjects who have not been hospitalised for more than 1 day for wLRI | 18 Months
  The proportion of subjects who have not been hospitalised for more than 1 day for wLRI during the Treatment period, during the Observational period, and during the whole study period will be assessed.

OTHER OUTCOMES:
Number of subjects with adverse events and serious adverse event | 18 Months
  The safety of short- and long-term treatment with OM-85 vs. placebo in children aged between 6 months and 5 years with recurrent RTIs associated with wLRI during the Treatment period and during the Observational period will be assessed.

CONTACTS AND LOCATIONS:
Locations (42):
- Germany (9):
  - Ludwig Maximilians Universität München, München, Bavaria
  - Clinical Research & Healthcare GmbH, Schönau am Königssee, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - St. Josef-Hospital, Bochum, North Rhine-Westphalia
  - University Hospital Cologne AöR, Cologne, North Rhine-Westphalia
  - Ev. Krankenhaus Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Praxis Köllges, Mönchengladbach, North Rhine-Westphalia
  - Marien-Hospital Wesel gGmbH, Wesel, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck, Schleswig-Holstein
- Hungary (6):
  - Aranyklinika Kft, Szeged, Csongrád megye
  - Dr. Kenessey Albert Korhaz-Rendelointezet, Balassagyarmat
  - Semmelweis Egyetem I.sz. Gyermekgyogyaszati Klinika, Budapest
  - Heim Pal Orszagos Gyermekgyogyaszati Intezet, Budapest
  - Sanitas Diagnosztikai és Rehabilitációs Központ, Gyula
  - Futurenest Kft., Miskolc
- Italy (5):
  - Osp.Pediatr.Giov.XXIII,AOUC P.Bari, Bari
  - ASST Papa GiovanniXXIII,Mat.Inf.Ped, Bergamo
  - Azienda ospedalo universitaria, Parma
  - Universita degli Studi di Pavia - Fondazione IRCCS Policlini, Pavia
  - SO S.Chiara, AOU Pisana, Pisa
- Poland (12):
  - Malopolskie Centrum Alergologii, Krakow, Lesser Poland Voivodeship
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Spolka z o.o., Tarnów, Lesser Poland Voivodeship
  - Centrum Alergologii Specjalistyczna Przychodnia Alergologiczna, Lublin, Lublin Voivodeship
  - WWCOiT im. M. Kopernika w Lodzi, Osrodek Pediatryczny im. dr J.Korczaka, Lodz, Lódzkie
  - NZOZ E-Vita, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Czestochowa, Częstochowa, Silesian Voivodeship
  - NZLA Michalkowice - Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie, Silesian Voivodeship
  - Centrum Medyczne PROMED, Krakow
  - Podkarpacki Osrodek Pulmonologii i Alergologii Sp. z o.o., Rzeszów
  - Velocity Skierniewice Sp. z o.o., Skierniewice
  - Przychodnia Specjalistyczna Prosen-Med NZOZ, Warsaw
  - NSZOZ Puls - Med Anna Bogusz, Agnieszka Musielak Sp.J., Skarżysko-Kamienna, Świętokrzyskie Voivodeship
- Switzerland (4):
  - CHUV-Centre Hopitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Inselspital Bern Kinderklinik, Bern
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Universitaets-Kinderklinik - Kinderspital Zuerich, Zurich
- United Kingdom (6):
  - Brighton And Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Royal Hospital for Children and Young People, Edinburgh
  - Royal London Hospital, London
  - King's College Hospital, London
  - Royal Manchester Children's Hospital - Paediatrics - Paediatrics, Manchester
  - Nottingham University Hospitals NHS Trust - Queen's Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: No